CLINICAL TRIAL: NCT01314456
Title: 3D Recording of a Trans-rectal Prostate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Bnai Zion Medical Center (Other Government); Barzilai Medical Center (Other); Meir Medical Center (Other)
Responsible Party: Michael Cohen, MD, Urology, HaEmek Medical center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NaviGo- 01; 3D TRUS Bx recording
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer; Benign Prostatic Hyperplasia
Keywords: Prostate biopsy; Trans-rectal ultrasound; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NaviGo (Experimental): Video recording of a normal TRUS guided prostate biopsy with additional 2 , non invasive,electromagnetic sensors attached to the TRUS probe and the patient's back,- to allow for a 3D modeling of the prostate.
  Interventions: Device: NaviGo

INTERVENTIONS:
Device: NaviGo — Video recording of a normal TRUS guided prostate biopsy with additional 2 , non invasive,electromagnetic sensors attached to the TRUS probe and the patient's back,- to allow for a 3D modeling of the prostate.
  Other Names: 3D recording of a trans-rectal prostate biopsy

SUMMARY:
Prostate biopsy is performed by multiple consecutive biopsy needle insertion into the prostate gland under a trans-rectal ultrasound probe guidance.

Today, the performing physician navigates the needle using a momentary 2D ultrasound image (longitudinal and transverse B mode) without any record of the full prostate boundaries or previous biopsies' location.

This study's Objectives are to record the trans-rectal biopsy procedure including the initial scan and the needle biopsy location and to modulate a 3D model of the prostate with accurate display the locations of the various biopsies taken during the procedure.

DETAILED DESCRIPTION:
3D record of a trans-rectal prostate biopsy

Clinical Study Protocol Study no: NaviGo -01

Sponsor: UC-CARE. Apollo Bld. 3rd fl. Hi-Tech Park P.O.Box 67 Yokneam 20692 Israel Tel: 972-4-9097427 Fax:972-4-9937323

Feb. 2011 Version: 02

ABBREVIATIONS:

3D: 3 Dimensional 2D: 2 Dimensional TR: Trans-Rectal

1. PROTOCOL SUMMARY Title: 3D recording of a trans-rectal prostate biopsy Device: Navigo™

   Study Objectives: 1) To record the trans-rectal biopsy procedure including the initial scan and the needle biopsy location 2) To modulate a 3D model of the prostate and accurately display the locations of the various biopsies taken during the procedure

   Study Design: Open prospective study. Recruitment target: 50 patients

   Study Population: Patients undergoing trans-rectal prostate biopsy

   Study endpoint:

   Accurate 3D modelling of the prostate and the biopsy procedure

   Principal Investigator

   Co-operating Company and Sponsor: Dr. Michael Cohen

   UC-CARE. Yokneam, Israel
2. INTRODUCTION Prostate biopsy is performed by multiple consecutive biopsy needle insertion into the prostate gland under the trans-rectal ultrasound probe guidance. The needle is inserted through a designated needle guide on the ultrasound probe, through the rectum wall and into the prostate gland.

Today, the performing physician navigates the needle using a momentary 2D ultrasound image (longitudinal and transverse B mode) without any record of the full prostate boundaries or previous biopsies' location. By recording the procedure the Navigo™ system will generate and display in off-line an accurate 3D model of the prostate and position the biopsies taken in the prostatic volume.

3. OBJECTIVES AND RATIONALE 3.1 Study objectives

1) To record the trans-rectal biopsy procedure including the initial scan and the needle biopsy location 2) To modulate a 3D model of the prostate and accurately display the locations of the various biopsies taken during the procedure

3.2 Rationale

The Navigo™ system is a noninvasive system that allows the physician to accurately record the biopsy procedure without changing the imaging system, the biopsy routine or the techniques used today to scan and guide the biopsy needle insertion. The ability to create an accurate 3D model of the prostate and accurately position the biopsy needle location will allow the performing physician a more precise navigation and easier and more accurate biopsy within the prostate volume and enable a better analysis of the procedure and the pathological results, hence improved clinical outcomes with intended therapy or surveillance ( i.e.- prepare for follow-up biopsy procedure if needed).

4. DEVICE DESCRIPTION AND INTENDED USE The Navigo™ system is comprised of two main elements: a standard laptop computer with a digitizer input to record incoming video input (from the ultrasound system), and an electro-magnetic 3D tracking system. The 3D tracking system is connected via USB to the laptop computer, the transmitter is placed beneath the patient's mattress and two sensors are attached,- one to the ultrasound probe (at the base/ non invasive part of the probe) and the other to the patient's back.

The Navigo™ system tracks and records the location of the ultrasound probe and the incoming video from the ultrasound system. The patient's movement is recorded and compensated when the ultrasound images are placed with reference to each other. In post procedure, the physician defines the boundaries of the prostate on selected ultrasound images and a 3D model of the prostate is displayed with all recorded biopsy specimens' locations displayed in the prostatic volume. The physician will be able to examine in post analysis the scattering quality of the biopsy specimens in the prostatic volume and update the pathology results. The 3D model can be rotated, manipulated and displayed in the physician's preferable choice.

The Navigo™ system is intended to record and display in 3D the biopsy procedure of any patient undergoing a prostate trans-rectal biopsy. The Navigo™ system is intended to record all the data from the initial scan, the volume measurements, and the biopsy needle insertion. All the images are saved and can be reviewed in post analysis, the needle location can be updated according to the physician's marking on the recorded ultrasound image and the pathology results will be displayed in color on the 3D model.

5. METHODS AND PROCEDURES 5.1 Study Design

The study is an open prospective study

* Examination procedure:

  o The trans-rectal ultrasound guided prostate biopsy procedure will be conducted with no change what so ever from the currently conducted procedure.

  o The exceptions to the normal procedure is the addition of the flat transmitter under the patients mattress, the 2 external attached sensors and the recording of the procedure via the video-out put of the ultrasound using the Navigo™ system.

  o The 3D model will be compared with the recorded ultrasound images by the physician
* The recorded data will be processed off-line (post biopsy /off-line analysis).
* The analysis of the results will be completed in post procedure by the physician.

5.2 Trial Procedure

* A short one-time calibration of the Navigo™ system with the ultrasound system will be completed by a trained technician (UC-CARE's technician)
* The transmitter will be placed beneath the patient's mattress and the body sensor will be attached to the patients' back using a regular disposable medical sticker.
* The trans-rectal ultrasound probe will be held by the physician and controlled throughout the procedure according to the existing current biopsy protocol, without any alterations.
* The common ultrasound video output will be connected to the video input of the Navigo™ system
* Patient's identifications will be filled to allow proper post examination analysis
* Following the initial scan of the prostate and the volume measurements the Navigo™ system will record the data and store it for post analysis
* In the 3D biopsy screen a 3D model of the prostate will be displayed with record of all needle biopsy locations as recorded during the procedure.
* The pathology results can be loaded to the Navigo™ system and displayed on the 3D model

  6. SUBJECT POPULATION SELECTION 6.1 Inclusion Criteria

  • Eligibility -
* Age 18 years or older
* Planned for trans-rectal prostate biopsy
* Signed informed consent

6.2 Exclusion criteria

* Patient's unwilling to participate
* Patients with metal prosthetics

  7. POTENTIAL BENEFITS TO SUBJECTS No immediate benefits are expected to be gained by the subjects participating in the study as the 3D modeling and the display is completed post procedure. The procedure will be carried out exactly as it would have been without the Navigo™ system participating in the biopsy procedure. The post procedure 3D model display with the biopsy specimen's location may enable better data analysis.

  8. POTENTIAL RISKS TO SUBJECTS The Navigo™ system is a passive system that does not require any change in the procedure performed today. The various components do not come in direct contact with the patient or the physician and the computer and 3D tracking system are well within the required safety protocols.

The Navigo system has been approved by the CE. The 3D tracking system is approved by the FDA for medical use and is classified as Type CF which is the most stringent classification, being required for those applications where the applied part is in direct conductive contact with the heart or other applications as considered necessary. The 3D tracking system is also part of an approved Helsinki trial in Bnei-zion hospital (monitoring of the birth progress, trial initiated by Dr. Yoav Paltieli) Adverse effects are not expected according to the accumulated experience with the 3D tracking system. Similarly, the Navigo™ system is not expected to add to the procedure any pain or discomfort to the patients.

9. SUBJECT RECUITMENT Study population will be recruited from the pool of patients who are scheduled for trans-rectal biopsy procedure

10. DATA ANALYSIS

The data analysis will include the following steps:

• Post procedure display of the prostate's 3D model and the location of the various biopsy specimens taken during the procedure in the prostatic volume

• Comparison of the results with the physician analysis of the specimens location as derived from the images themselves

11. REFERENCE

1. Ultrasonography and biopsy of the prostate. Ramey et al., Chapter 92. Campbell-Walsh Urology. Elsevier 2007.
2. Prostate biopsies guided by three-dimensional real-time (4-D) transrectal ultrasonography on a phantom: comparative study versus two-dimensional transrectal ultrasound-guided biopsies. Long, Eur.Urol, 2007 Oct;52(4):1097-104.
3. Extended and saturation prostatic biopsy in the diagnosis and characterisation of prostate cancer: a critical analysis of the literature. Scattoni , Eur Urol. 2007 Nov;52(5):1309-22 .
4. Appropriate Patient Selection in the Focal Treatment of Prostate Cancer: The Role of Transperineal 3-Dimensional Pathologic Mapping of the Prostate-A 4-Year Experience. Barzell. Urology 70 ( suppl. 6a) dec. 2007
5. The lottery of conventional prostate biopsy. Andriole. Nat. Rev. urol. P-189 , V-6, Apr. 2009
6. Will focal therapy become a standard of care for men with localized prostate cacner? Ahmed. Nat. Clin.Pract. Oncol. 4(11)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Planned for trans-rectal prostate biopsy
* Signed informed consent

Exclusion Criteria:

* Patient's unwilling to participate
* Patients with metal prosthetics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Create 3D model of the prostate and accurately display the locations of the various biopsies taken during the procedure | Post procedure ( off-line ) within a 3-5 working days

CONTACTS AND LOCATIONS:
Overall Officials: Boris Yudkevich, MD, Study Director — HaEmek Medical Center, Israel; Genady Zelichenko, MD, Study Director — HaEmek Medical Center, Israel; Ilan Leibovich, MD, Principal Investigator — Meir Medical center, Israel; Giora Tikotchinsky, MD, Study Director — Meir medical center, Israel; Moshe Shalev, MD, Study Director — Meir medical center, Israel; Ofer Nativ, Prof., MD, Principal Investigator — Bnei-Zion medical center, Israel; Shmuel Cytron, MD, Principal Investigator — Barzilai medical center, Israel; Michael Cohen, MD, Principal Investigator — HaEmek Medical Center, Israel
Locations (1):
- Dept. of urology , HaEmek medical center, Afula, Israel